CLINICAL TRIAL: NCT00000775
Title: A Phase I Safety and Immunogenicity Trial of UBI SynVac (HIV-1 MN Octameric V3 Peptide Vaccine)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Masking: Double | Purpose: Prevention
Other Study IDs: AVEG 011
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-10

CONDITIONS: HIV Infections
Keywords: Vaccines, Synthetic; HIV-1; HIV Envelope Protein gp120; AIDS Vaccines; HIV Seronegativity; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Biological: rgp120/HIV-1MN Monovalent Octameric V3 Peptide Vaccine

SUMMARY:
To determine the safety, immunogenicity, and optimal dose of rgp120/HIV-1MN octameric V3 peptide vaccine (SynVac) in healthy volunteers.

It is likely that the ultimate control of AIDS will depend on the development of safe and effective vaccines against HIV-1. SynVac is a synthetic candidate vaccine based on eight V3-derived peptides attached to a heptalysyl core to form radial octamers. In animal studies, the vaccine appears safe and demonstrates the capability for producing immune responses.

DETAILED DESCRIPTION:
It is likely that the ultimate control of AIDS will depend on the development of safe and effective vaccines against HIV-1. SynVac is a synthetic candidate vaccine based on eight V3-derived peptides attached to a heptalysyl core to form radial octamers. In animal studies, the vaccine appears safe and demonstrates the capability for producing immune responses.

Twelve volunteers are entered at one of three dose levels of SynVac. At each dose level, 10 volunteers receive vaccine and two receive placebo. At least eight volunteers at each dose level must be monitored for 1 week before subsequent volunteers are entered at the next higher level. Intramuscular injections are given on day 0, 28, and 168. Approximately 12 clinic visits are required.

ELIGIBILITY:
Inclusion Criteria

Subjects must have:

* Normal history and physical exam.
* Negative for HIV by ELISA within 6 weeks of immunization.
* CD4 count >= 400 cells/mm3.
* Normal urinalysis.

Exclusion Criteria

Co-existing Condition:

Subjects with the following conditions are excluded:

* Medical or psychiatric condition or occupational responsibilities that preclude compliance.
* Active syphilis (volunteers are eligible if serology is documented to be a false positive or due to a remote (> 6 months) treated infection).
* Active tuberculosis (volunteers with a positive PPD and normal chest x-ray showing no evidence of TB and not requiring INH therapy are eligible).
* Hepatitis B surface antigenemia.

Subjects with the following prior conditions are excluded:

* History of immunodeficiency, chronic illness, autoimmune disease, or use of immunosuppressive medications.
* History of anaphylaxis or other serious adverse reactions to vaccines.

Prior Medication:

Excluded:

* Live attenuated vaccines within the past 60 days. NOTE: Medically indicated subunit or killed vaccines (e.g., influenza, pneumococcal) are permitted if received at least 2 weeks prior to first immunization.
* Experimental agents within the past 30 days.
* Prior HIV vaccines.

Prior Treatment:

Excluded:

* Blood products or immunoglobulin within the past 6 months.

Identifiable high-risk behavior for HIV infection, including history of injection drug use within the last 12 months prior to enrollment and higher or intermediate risk sexual behavior.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40

CONTACTS AND LOCATIONS:
Overall Officials: Gorse G, Study Chair
Locations (2):
- United States (2):
  - St Louis Univ School of Medicine, St Louis, Missouri
  - Univ of Rochester Med Ctr, Rochester, New York

REFERENCES:
- [Background] Gorse GJ, Keefer MC, Belshe RB, Matthews TJ, Forrest BD, Hsieh RH, Koff WC, Hanson CV, Dolin R, Weinhold KJ, Frey SE, Ketter N, Fast PE. A dose-ranging study of a prototype synthetic HIV-1MN V3 branched peptide vaccine. The National Institute of Allergy and Infectious Diseases AIDS Vaccine Evaluation Group. J Infect Dis. 1996 Feb;173(2):330-9. doi: 10.1093/infdis/173.2.330. PMID 8568293